Growth Mindset Psychoeducation for Modifiable Risk Factors for CMD NCT03707522 05/31/2018

# University of Nevada, Reno Social Behavioral or Educational Research Consent Form

Title of Study: Freshmen Wellness Principal Investigator: Anthony Papa, PhD

(775) 682-8666

Co-Investigators / Martha Zimmermann, MA

Study Contact: (775) 636-8067

mzimmermann@nevada.unr.edu

**Study ID Number:** 1240550-1

Sponsor: N/A

#### Introduction

You are being invited to participate in a research study. Before you agree to be in the study, read this form carefully. It explains why we are doing the study; and the procedures, risks, discomforts, benefits and precautions involved.

At any time, you may ask one of the researchers to explain anything about the study that you do not understand.

It's important you are completely truthful about your eligibility to be in this study. If you are not truthful, you may be harmed by being in the study.

You do not have to be in this study. Your participation is voluntary. If you do not agree to participate, you will receive the **education** you would have received if the study was not taking place.

Take as much time as you need to decide. If you agree now but change your mind, you may quit the study at any time. Just let one of the researchers know you do not want to continue.

#### Why are we doing this study?

We are doing this study to find out more about the impact of learning about about mental health on mental health and quality of life. Benefits of research cannot be guaranteed but we hope to learn more about the impact of learning more about mental health on wellness and health.

## Why are we asking you to be in this study?

We are asking you to be in this study because you indicated that you are older than 18, an English speaker, and that you are an incoming UNR freshmen.

# How many people will be in this study?

We expect to enroll 500 participants at the University of Nevada, Reno.

Page 1 of 4

05/31/2018

# What will you be asked to do if you agree to be in the study?

If you agree to be in this study you will be asked to answer some questions about yourself, including your experience in the last two weeks. You will also be asked about some health habits and behaviors that you engage in. You will then be asked to read an article and some information about mental health and respond to some brief questions about what you have read.

You will be contacted during the Fall semester for a follow-up questionnaire regarding emotional experiences and health behaviors.

#### How long will you be in the study?

The study will take about 45 minutes of your time, 30 minutes now and 15 minutes at a follow up date in the Fall. You'll participate for about 2-3 months.

# What are your choices if you do not volunteer to be in this research study?

If you decide not to be in the study, you may discontinue your participation at any time.

#### What if you agree to be in the study now, but change your mind later?

You do not have to stay in the study. You may withdraw from the study at any time by informing a member of the research team that you would like to withdraw from the study.

## What if the study changes while you are in it?

If anything about the study changes or if we want to use your information in a different way, we will tell you and ask if you if you want to stay in the study. We will also tell you about any important new information that may affect your willingness to stay in the study.

### Is there any way being in this study could be bad for you?

We do not anticipate any risks involved in participating in this study. However, if you feel uncomfortable answering any questions, you can withdraw from the study at any time.

#### What happens if you become injured because of your participation in the study?

We do not anticipate any risks involved in participating in this study

#### Will being in this study help you in any way?

We cannot promise you will benefit from being in this study but you may learn some new information about mental health and strategies for promoting mental wellness.

#### Who will pay for the costs of your participation in this research study?

No costs are associated with participation in this study.

#### Will you be paid for being in this study?

You will not receive any payment for being this study. If you complete the follow-up questionnaire in the Fall, you will be compensated 1 SONA credits. This may count for course credit if you are in a course that allows for the use of SONA credits.

Page 2 of 4 05/31/2018

# Who will know that you are in in this study and who will have access to the information we collect about you?

The researchers, the University of Nevada, Reno Institutional Review Board, and US Department of Health and Human Services (DHHS) will have access to your study records. A description of this clinical trial will be available on http://www.ClinicalTrials.gov as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

#### How will we protect your private information and the information we collect about you?

We will treat your identity with professional standards of confidentiality and protect your private information to the extent allowed by law. We will do this by giving your information a participant ID that is not associated with your name or any other identifying information. Any information containing your name or contact information will be destroyed upon completion of the study.

We may publish the information from this study in journals or present it at research conferences. If we do, we will not use your name or other identifying information. No personal identifying information will be included in this database. We will not use your name or other information that could identify you in any reports or publications that result from this study.

Do the researchers have monetary interests tied to this study? No.

# Who can you contact if you have questions about the study or want to report an injury?

At any time, if you have questions about this study or wish to report an injury that may be related to your participation in this study, contact Anthony Papa, PhD at (775) 682-8666 or Martha Zimmermann at (775) 636-8067.

Who can you contact if you want to discuss a problem or complaint about the research or ask about your rights as a research participant?

You may discuss a problem or complaint or ask about your rights as a research participant by calling the University of Nevada, Reno Research Integrity Office at (775) 327-2368. You may also use the online *Contact the Research Integrity Office* form available from the *Contact Us* page of the University's Research Integrity Office website.

# Agreement to be in study

| If you agree to participate in this study, you must sign this consent form. We will give you a copy of the form to keep. | |
|---|---|
| Participant's Name Printed | |
| Signature of Participant | Date |
| Signature of Person Obtaining Consent | Date |